CLINICAL TRIAL: NCT05041517
Title: Brief Online Training (BOLT) for Routine Outcome Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Lyon, Associate Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 52550; R34MH109605 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Mental Health Issue; Adoption of Measurement-Based Care (MBC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No intervention
- BOLT + 1 PTC (Experimental): BOLT Training + 1 PTC Call
  Interventions: Behavioral: BOLT + PTC
- BOLT + 2 PTC (Experimental): BOLT Training + 2 PTC Calls
  Interventions: Behavioral: BOLT + PTC
- BOLT + 4 PTC (Experimental): BOLT Training + 4 PTC Calls
  Interventions: Behavioral: BOLT + PTC

INTERVENTIONS:
Behavioral: BOLT + PTC — BOLT is a Brief Online Training (BOLT) for Measurement-Based Care (MBC). Participants in the BOLT condition were subsequently randomized into varying amounts of post-training consultation (PTC).
  Arms: BOLT + 1 PTC; BOLT + 2 PTC; BOLT + 4 PTC

SUMMARY:
The goal of this project is to improve school-based services by developing and testing an online training and consultation system to facilitate the use of measurement-based care (also known and referenced in original grant as routine outcome monitoring). Measurement-based care (MBC) is the target intervention because it is an EBP with extensive empirical support for its ability to improve mental health service outcomes and is a feasible and cost-effective option. Following the iterative development of the BOLT training and consultation package (phases 1-4), the investigators will conduct a randomized control pilot trial (phase 5) to test the (1) impact of the package on MBC knowledge, attitudes and use, (2) impact of varying degrees of consultation dosage on weekly assessments of MBC use, and (3) moderators and mechanisms of impact.

DETAILED DESCRIPTION:
In the US, although roughly one in five children experiences a mental health problem severe enough to warrant diagnosis and intervention, most lack access to needed services. Schools offer opportunities to improve service access, but school mental health clinicians are unlikely to deliver high-quality evidence-based practices (EBP). Multiple barriers interfere with clinicians receiving adequate training and support for EBP, including limited time and scarce training resources. The goal of this project is to improve school-based services by developing and testing an online training and consultation system to facilitate the use of measurement-based care (MBC). MBC is the target intervention because it is an EBP with extensive empirical support for its ability to improve mental health service outcomes and is a feasible and cost-effective option.

The larger study was conducted in phases to address study aims (this clinical trial record reflects Aim 3/Phase 5):

* AIM 1: Phases 1 and 2. Develop the Brief On-Line Training (BOLT) for Measurement-Based Care training through prototyping and continuous user testing. The goal is to optimize BOLT's impact on system usability and clinician gains in MBC knowledge and attitudes.
* AIM 2: Phases 3 and 4. Develop the BOLT post-training consultation procedures to optimize effective consultation.
* AIM 3: Phase 5. Test BOLT by conducting a randomized controlled pilot trial of the full BOLT training/consultation package to test (1) its impact on MBC knowledge, attitudes, and use; (2) the impact of varying degrees of consultation dosage on weekly assessments of MBC use; and (3) moderators and mechanisms of impact: (a) system usability, (b) clinician knowledge and attitudes gain, (c) experience of collaboration, and (d) responsiveness of consultation.

During the final year (i.e., phase 5), participants include a sample of 75 clinicians, recruited from national email listservs in order to most closely approximate how clinicians tend to discover and engage in online training opportunities. Participants complete an initial online survey about their use of MBC in practice and are randomly assigned to participate in one of two study conditions: the BOLT condition (training and consultation) or a Control condition (no training and no consultation). Participants in the BOLT condition complete a self-paced Brief Online Training (BOLT) for Measurement-Based Care (MBC), are asked to begin to use MBC with their caseloads, and are then randomly assigned to one of three different consultation groups receiving 2 weeks, 4 weeks or 8 weeks of consultation. Participation in a consultation group includes participating in biweekly group phone consultations and posting weekly assignments on an online consultation discussion board about their use of MBC in practice. Participants in all BOLT groups and the Control condition complete weekly online surveys for the full 32 weeks of data collection.

ELIGIBILITY:
Inclusion Criteria:

* Between 22-80 years of age
* Employed as a School-Based Mental Health provider
* Must routinely provide individual-level interventions or therapy to students and spend >50% of their time providing services in schools

Exclusion Criteria:

* Being younger than 22 or older than 80
* Not being employed as a School-Based Mental Health provider
* Don't provide individual-level interventions or therapy to students nor spend >50% of their time providing services in schools.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Current Assessment Practice Evaluation - Revised (CAPER) - Change of use of MBC | Baseline, Weeks 2-32
  The CAPER includes the original four-item CAPE measure plus three new items to assess use of individualized assessment. It assesses clinician self-reported use of the full range of MBC practices including administration of individualized/standardized assessments at different points during treatment, client feedback on assessment results, and using assessment results to inform treatment. All items are scored on a 1-4 scale, with anchors signifying percent of clients they used the practice with: 1 = None (0%), 2 = Some (1-39%), 3 = Half (40-60%), 4 = Most (61-100%).
Monitoring & Feedback Attitudes Scale (MFAS) - Change of attitudes about MBC use | Baseline, Weeks: 2,4,6,8,10,16,20,24,28,32
  The purpose of this measure is to collect information on attitudes on routine progress monitoring (or measurement-based care). Monitoring and Feedback Attitudes Scale (MFA; Jensen-Doss, Becker, Smith, Lyon, Lewis, Stanick, & Hawley, 2018) responses range from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). The MFA has two subscales: (1) Benefit (i.e., facilitating collaboration with clients) and (2) Harm (i.e., harmful for therapeutic alliance, misuse by administrators).
MBC Knowledge Questionnaire (MBCKQ) - Change of knowledge about MBC | Baseline, Weeks: 2,4,6,8,10,16,20,24,28,32
  The purpose of this questionnaire is to measure MBC knowledge. The 28-item, multiple-choice MBCKQ was iteratively developed based on the key content and learning objectives of the MBC training modules.
Routine-Outcome Monitoring Skill - Change of skill of MBC use | Baseline, Weeks: 2,4,6,8,10,16,20,24,28,32
  The purpose of this measure is to collect information on clinician familiarity and use of routine outcome monitoring (both individualized and standardized assessment tools). Items address selection of clients for administration as well as tool selection, administration, scoring, interpretation, integration into treatment, feedback, and progress monitoring. In previous samples, the scale had good internal consistency (Cronbach's α = .85). Responses are ratings about skill level and practice, ranging from 1 (''Minimal'') to 5 (''Advanced''). Items are averaged to create a total assessment skill score.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lyon, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Lyon AR, Liu FF, Connors EH, King KM, Coifman JI, Cook H, McRee E, Ludwig K, Law A, Dorsey S, McCauley E. How low can you go? Examining the effects of brief online training and post-training consultation dose on implementation mechanisms and outcomes for measurement-based care. Implement Sci Commun. 2022 Jul 22;3(1):79. doi: 10.1186/s43058-022-00325-y. PMID 35869500